CLINICAL TRIAL: NCT01173250
Title: Is Diverting Ileostomy Necessary in Stapled Ileoanal Pouch?
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mansoura University (Other)
Other Study IDs: 251068
Record Dates: First submitted 2010-07-30; First posted 2010-08-02 (Estimated); Last update posted 2010-08-16 (Estimated); Status verified 2010-10

CONDITIONS: Ulcerative Colitis; Familial Adenomatous Polyposis
Keywords: total proctocolectomy with ileal pouch anal anastomosis with and without ileostomy
MeSH Terms: conditions — Colitis, Ulcerative; Adenomatous Polyposis Coli

ARMS (2):
- stapled ileoanal pouch without diverting ileostomy (Active Comparator)
  Interventions: Procedure: omitting diverting ileostomy
- stapled ileoanal pouch with diverting ileostomy (Placebo Comparator)
  Interventions: Procedure: adding diverting ileostomy

INTERVENTIONS:
Procedure: adding diverting ileostomy
  Arms: stapled ileoanal pouch with diverting ileostomy
Procedure: omitting diverting ileostomy
  Arms: stapled ileoanal pouch without diverting ileostomy

SUMMARY:
Total proctocolectomy with ileal pouch anal anastomosis is the first choice surgical operation for management of ulcerative colitis and familial adenomatous polyposis. The addition of diverting ileostomy may reduce septic complications. In this randomized study the investigators compare two groups of patients with stapled ileoanal pouch one of them had diverting ileostomy and in the other this step is omitted.

ELIGIBILITY:
Inclusion Criteria:

* patients having total proctocolectomy with ileal pouch anal anastomosis.

Exclusion Criteria:

* hypoalbuminemia
* prolonged steroid use
* anemia
* anastomosis under tension
* leak with air test
* bleeding
* poor vascular supply of anastomosis

Sex: All
Age Groups: Child, Adult, Older Adult